CLINICAL TRIAL: NCT05347030
Title: Acupuncture for Impaired Glucose Tolerance in Overweight/Obese Population: a Multi-center Randomized Controlled Trial
Brief Title: Acupuncture for Impaired Glucose Tolerance in Overweight/Obese Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yan Yan (Other)
Responsible Party: Sponsor-Investigator, Yan Yan, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-021-KY-01
Record Dates: First submitted 2022-04-18; First posted 2022-04-26 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Impaired Glucose Tolerance; Overweight; Obese; Prediabetic State
Keywords: impaired glucose tolerance; overweight; obese; Prediabetic State; acupuncture; randomized controlled trial
MeSH Terms: conditions — Glucose Intolerance; Overweight; Obesity; Prediabetic State | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Group (Experimental): The acupuncture points are: EX-B3, BL18, BL20, BL21, GV20, GV29, LI11, CV12, CV10, ST25, CV6, CV4, ST40, SP6.
  After piercing 15-35mm into the skin, the needles will be gently rotated and lifted three times to achieve a sense of sourness, distention, and heaviness (de qi). For EX-B3, BL18, BL20, and BL21, withdrawn afterward immediately. For GV20, GV29, LI11, CV12, CV10, ST25, CV6, CV4, ST40 and SP6, The needles will be maintained for 30 minutes.
  Interventions: Other: Acupuncture
- Sham Acupuncture Group (Sham Comparator): sham acupoints are located at a horizontal distance of 20 mm to those points used in the acupuncture group, and no manipulation was carried out after piercing the skin for 1-2mm to avoid de-qi sensation.
  For sham EX-B3, BL18, BL20, and BL21, withdraw immediately after piercing. For sham GV20, GV29, LI11, CV12, CV10, ST25, CV6, CV4, ST40 and SP6, The needles will be maintained for 30 minutes after puncture.
  Interventions: Other: Sham Acupuncture

INTERVENTIONS:
Other: Acupuncture — During the 12-week treatment, acupuncture will be administrated 3 times a week (once every other day) in the first 6 weeks, and twice a week in the last 6 weeks (with an interval of 2-3 days). Each treatment session will last 30 minutes.
  Arms: Acupuncture Group
Other: Sham Acupuncture — During the 12-week treatment, Sham Acupuncture will be administrated 3 times a week (once every other day) in the first 6 weeks, and twice a week in the last 6 weeks (with an interval of 2-3 days). Each treatment session will last 30 minutes.
  Arms: Sham Acupuncture Group

SUMMARY:
This is a prospective, multicenter, parallel-group, participants- and assessors-blinded randomized trial aiming to evaluate the effectiveness and safety of acupuncture in improving glucose metabolism for overweight/obese Participants with IGT, in comparison with sham acupuncture.

DETAILED DESCRIPTION:
The trial will be conducted at three hospitals in China. 196 eligible subjects will be randomly assigned (1:1) to the acupuncture or sham acupuncture group to receive either 30-session acupuncture/sham acupuncture treatment over 12 weeks based on lifestyle intervention and 24-week follow-up. The primary outcome is the change in the value of 2-hour blood glucose (2hPG) from baseline at the end of the 12-week treatment. Additionally, compliance, blinding, and safety will also be assessed. All statistical tests will be performed using a two-sided test, a p-value of less than 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. those who meet the diagnostic criteria of overweight/obesity and IGT:

   ①IGT: fasting blood glucose (PG) is lower than 7.0mmol/L, and 2-hour blood glucose (2hPG) after oral 75g glucose tolerance test (OGTT) is between 7.8~11.1mmol/L.

   ②overweight: 24.0 < BMI ≤ 27.9, obesity: BMI ≥ 28.0, or BMI ≤24.0 but Waist Circumference ≥85 cm (male) /≥80 cm(female).
2. 18-60 years old;
3. those who can appropriately describe their wishes, voluntarily fill in the informed consent form and agree to participate in clinical trials.

Exclusion Criteria:

1. obesity secondary to heredity, drugs, and diseases;
2. those who have received weight-loss treatment including acupuncture and drugs in the past 3 months;
3. those who have taken drugs that have known effects on body weight or appetite in the past 3 months, such as corticosteroids, antidepressants, non-selective antihistamines in vivo, nicotine substitutes, etc;
4. IGT is caused by abnormal thyroid function, endocrine tumors, extensive liver damage;
5. abnormal glucose tolerance caused by thiazide diuretics, β-blockers, nicotinic acid drugs, quinolones, calcineurin inhibitors, interferon-alpha, etc;
6. received antidiabetic medicines in the past 3 months；
7. participants with serious primary diseases such as heart, lung, brain, liver, or hematopoietic system diseases, progressive malignant tumor, or other serious consumptive diseases;
8. Participants with cognitive impairment and severe mental illness;
9. participants with blood coagulation dysfunction, and scare of needles；
10. pregnant, breastfeeding, or planning to conceive within 37 weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 196 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in the value of 2-hour blood glucose from baseline at the end of the 12-week treatment | week 12
  The 2-hour blood glucose is the value of intravenous plasma glucose measured by oral 75g glucose tolerance test, which is usually used to diagnose impaired glucose tolerance and observe glucose metabolism.

SECONDARY OUTCOMES:
The change in the value of 2-hour blood glucose from baseline | weeks 24 and 36
  The 2-hour blood glucose is the value of intravenous plasma glucose measured by oral 75g glucose tolerance test, which is usually used to diagnose impaired glucose tolerance and observe glucose metabolism.
The proportion of participants whose 2-hour blood glucose dropped to normal from baseline | weeks 12, 24 and 36
  The 2-hour blood glucose is the value of intravenous plasma glucose measured by oral 75g glucose tolerance test, which is usually used to diagnose impaired glucose tolerance and observe glucose metabolism.
The proportion of participants with at least 5% reductions in body weight from baseline | weeks 4, 8, 12, 16, 24 and 36
  The body weight will be reported in kg.
The change from baseline of body mass index | weeks 4, 8, 12, 16, 24 and 36
  The body mass index is a figure obtained by dividing body weight by the square of height, in kilograms per meter^2. It is a universal indicator used in the world to measure the degree of obesity.
The change from baseline of fasting plasma glucose | weeks 12, 24 and 36
  The fasting plasma glucose is measured by oral 75g glucose tolerance test, which is usually used to diagnose impaired glucose tolerance and observe glucose metabolism.
The change from baseline of Fasting serum insulin | weeks 12, 24 and 36
  The fasting serum insulin is measured by oral 75g glucose tolerance test, which was used to diagnose impaired glucose tolerance and observe glucose metabolism.
The change from baseline of Homeostasis model assessment-insulin resistance | weeks 12, 24 and 36
  Homeostasis model assessment-insulin resistance index (HOMA-IR): a mathematical model reflecting the interaction of glucose and insulin in different organs (including pancreas, liver, and surrounding tissues). It was first proposed by Matthews in 1985. Insulin resistance (HOMA-R) and islet β cell function (HOMA- β) were evaluated by fasting blood glucose value (FPG) and fasting serum islet level (FINS). The calculation method is HOMA-IR=FPG × FINS/225;HOMA- β = 20 × FINS/ (FPG-3.5). The FPG unit is mmol/L, FINS μ U/ml, and the coefficient 225is the correction factor, which refers to the blood glucose level of 5 μ U / ml plasma insulin corresponding to 45mmol/L in normal/ideal individuals.
The change from baseline of Waist-to-Hip Ratio | weeks 4, 8, 12, 16, 24 and 36
  Waist-to-Hip Ratio(WHR): the ratio of waist to hip circumference. It is an important measure for the diagnosis of central adiposity.
  To measure waist circumference, locate the upper hip bone and the top of the right iliac crest. Place a measuring tape in a horizontal plane around the abdomen at the level of the iliac crest. To measure hip circumference, place the measuring tape on the horizontal plane and place it at the maximum extension of the hip.
  Before reading the tape measure, ensure that the tape is snug, but does not compress the skin, and is parallel to the floor. The measurement is made at the end of a normal expiration.
The change from baseline in the SNAQ scores | weeks 4, 8, 12, 16, 24 and 36
  SNAQ=simple appetite questionnaire. SNAQ is a short and simple appetite assessment tool that can predict weight loss in adults. It measures the amount of food per meal, the number of meals per day, and the taste of the food. It consists of four items, each with five grades, with the total score ranging from 4 to 20 points. Lower scores indicate deterioration in appetite.
The change from baseline in the IWQOL-Lite scale scores | weeks 4, 8, 12, 16, 24 and 36
  IWQOL-Lite=Impact of Weight on Quality Of Life. IWQOL-Lite is an international scale used to measure an individual's health-related quality of life. A total of 31 questions are divided into five subscales: 11 questions concerning physical function, 7 concerning self-esteem, 4 concerning sex life, 5 concerning public pressure, and 4 concerning work. The score of each question is divided into five grades, with 5 representing always, 4 often, 3 sometimes, 2 rarely and 1 never. The total score of the questionnaire is 155, with a higher score indicating a worse quality of life.
The change from baseline of TC, TG, LDL-C, and HDL-C | weeks 12, 24 and 36
  TC=Serum total cholesterol, TG=triglyceride, LDL-C=Low-Density Lipoprotein Cholesterol, HDL-C=High-Density Lipoprotein Cholesterol. They are important indicators to evaluate the metabolism of blood lipids in the human body, all of which will be reported in mmol/L.
The change from baseline of blood pressure | weeks 12, 24 and 36
  The blood pressure is measured by an OMRON upper arm blood pressure electronic sphygmomanometer. Before blood pressure measurement, subjects are required to sit still for five minutes, relax the whole body and take three slow deep breaths; during blood pressure measurement, subjects must keep their wrists still and placed at the same level as the heart. Keep calm and do not speak during the measurement. The blood pressure was measured 2 times and the average blood pressure was taken as the actual blood pressure.

OTHER OUTCOMES:
Expectation assessment | baseline
  Participants will be asked "Do you think acupuncture will be effective for treating the illness?" and "Do you think acupuncture will be effective for controlling weight and improving glucose?" The response options will be "Ineffective", "the effect is not good", "uncertain", "has some effect", or "very effective".
Blinding assessment | week 12
  Participants will be told that insertion is deeper in traditional acupuncture group and shallower in modern acupuncture group. After treatments finished, they will be asked "Do you think you have received traditional acupuncture in the past weeks?", the answers are "Yes", "No" or "Unclear".
Compliance assessment of acupuncture | week 12
  compliance = (the times the Participant has received acupuncture/ the total times the Participant should receive acupuncture ) × 100% the criterion of good compliance was that the Participants had received more than 80% of treatment (including 80%).
Compliance assessment of life modification | weeks 4, 8, 12, 16, 24 and 36
  The patient's lifestyle adjustment diary card, dietary change table, dietary compliance questionnaire, and exercise compliance scale were selected to evaluate the compliance of life modification.
Incidence of Adverse Events | week 0 to 36
  Acupuncture-related adverse events(such as broken needles, hematoma, infection, etc.) and other unexpected adverse events(such as colds, falls, etc.), including their severity and possible relationship with interventions, will be recorded in detail in the patient-recorded adverse event table and the evaluator-recorded adverse event table throughout the study period. The incidence of adverse events in the two groups will be calculated at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Yan, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, Beijing, China

REFERENCES:
- [Derived] Yan Y, Sun Y, Wang X, Zhu L, Chen Y, Liu Z. Acupuncture for Impaired Glucose Tolerance in People With Obesity: A Protocol for a Multicenter Randomized Controlled Trial. Front Med (Lausanne). 2022 Jul 12;9:932102. doi: 10.3389/fmed.2022.932102. eCollection 2022. PMID 35903320